CLINICAL TRIAL: NCT06890962
Title: The Effect of Citicoline and Caffeine Dose in a Commercial Energy Drink on Cognitive Performance, Energy Expenditure and Fat Oxidation in Young Adults
Brief Title: Citicoline Dose on Energy Drink Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathaniel Jenkins (Other)
Collaborators: Woodbolt Distribution (Unknown)
Responsible Party: Sponsor-Investigator, Nathaniel Jenkins, Assistant Professor, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 202302574
Record Dates: First submitted 2024-06-03; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Performance; Gaming Performance; Blood Pressure; Heart Rate; Mood

STUDY DESIGN:
Intervention Model Description: 4 condition, randomized cross-over with 3-7 day washout between conditions
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Energy Drink (Active Comparator): C4 Smart Energy, 1 can, administered acutely
  Interventions: Dietary Supplement: Energy drink consumption
- Reduced Citicoline Energy Drink (Experimental): C4 Smart Energy Reduced Citicoline, 1 can, administered acutely
  Interventions: Dietary Supplement: Energy drink consumption
- Reduced Citicoline and Caffeine Energy Drink (Experimental): C4 Smart Energy Reduced Citicoline and Caffeine, 1 can, administered acutely
  Interventions: Dietary Supplement: Energy drink consumption
- Placebo (Placebo Comparator): Placebo Drink devoid of active ingredients, 1 can, administered acutely
  Interventions: Dietary Supplement: Energy drink consumption

INTERVENTIONS:
Dietary Supplement: Energy drink consumption — Participants will consume an energy drink (or placebo) and then undergo experimental testing after a 40 minute rest period following drink consumption.

SUMMARY:
The purpose of this study is to determine how the doses of cognitive-enhancing ingredients such as citicoline and caffeine effect the efficacy of acute energy drink consumption for improving cognitive performance (primary outcome), gaming performance, mood, energy expenditure, and fat oxidation. This study will utilize an In vivo acute response, randomized, double-blind, placebo controlled, cross-over trial study design. Participants will complete consent, complete screening, and then undergo familiarization and complete four experimental study visits. In brief, participants will consume a commercially available energy drink specifically formulated to improve cognitive performance with the standard dose of Cognizin, a reduced dose of Cognizin, a reduced dose of caffeine and Cognizin, or a placebo (water, which will be carbonated, matched for flavor, mouthfeel, etc.), then complete a battery of computer-based cognitive performance test, tasks in a video game (Tetris) to assess video game performance, have their resting metabolism analyzed, and then assessments of mood. Following a 1-week washout period, participants will return and consume one of the four remaining beverages and complete the same tasks. They will participate in four experimental visits, each time consuming a different beverage until they have consumed all beverages and completed all necessary tasks.

Question(s) and Hypotheses (stated in null) Q: Does acute consumption of a new formulations (reduced active ingredients [citicoline and caffeine]) of a commercially available energy drink elicit similar improvements in cognitive performance, mood, energy expenditure and fat oxidation in young adults than the standard, currently marketed dose to formulation?

H1: Acute consumption of the commercially available energy drink with standard dosing will improve cognitive performance compared to the reduced dose beverages and the placebo.

H2: Acute consumption of the commercially available energy drink with standard dosing will improve gaming (Tetris) performance compared to the reduced dose beverages and the placebo.

H3: Acute consumption of the commercially available energy drink with standard dosing will improve mood compared to the reduced dose beverages and the placebo.

H4: Acute consumption of a commercially available energy drink with standard dosing will increase energy expenditure and fat oxidation compared to the reduced dose beverages and the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Fitness: Healthy, recreationally trained (>2 d/wk physical activity)
* BMI: (<30kg/m2) or BF <25% (M) and <32% (F)

Exclusion Criteria:

* <1 hr/wk playing video games
* >=21 servings of >=170.5 mL (or >=6 fl oz) caffeine beverages per week [(PMID: 33525438)]
* Injury or illness
* Habitual nicotine or cannabis use
* Use of prescription ADD/ADHD, anti-depressant, or other central acting medication, or previously diagnosed ADD/ADHD, clinical depression, or other mental health condition
* Use of prescription, OTC, or dietary supplements to support sleep, or having been diagnosed with a clinical sleep condition
* Current or prior chronic (>6 mo) illicit drug or alcohol abuse
* Clinically diagnosed with, or taking medication for a cardiometabolic disease or disorder (e.g., Pre-diabetes, Type II diabetes, high blood pressure, chronic kidney disease, cardiovascular disease, obesity, etc.)
* Clinically diagnosed digestive disorder or sensitivity, or regular use of OTC or dietary supplements to support gastrointestinal pain or discomfort
* Competitive athlete
* Failure to comply with the controls and conditions of this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Executive Function | 60 minutes post-drink consumption
  How well a subject recognizes rules, categories, and manages or navigates rapid decision making. Assessed as Shifting Attention Task (SAT) Correct Responses - SAT Errors.
Resting Fat Oxidation | 50 minutes post-drink consumption
  Resting fat oxidation (g/min) will be quantified from resting, fasted analyses of pulmonary gas exchange.
Video Game Performance | 90 minutes post-drink consumption
  Performance in the two-dimensional visuospatial game Tetris. Participants will be given four minutes of play time on Marathon mode and instructed to maximize the score (points) displayed on the screen. The total score at the end of play time will be recorded.

SECONDARY OUTCOMES:
Sustained Attention | 60 minutes post-drink consumption
  Measure of how well a subject can direct and focus cognitive activity on specific stimuli. Assessed using the 4-part Continuous Performance Test, which requires the subject to respond to the target stimulus "B" but not to any other letter. Stimuli are presented at random and the subject responds by pressing the SPACE BAR. Sustained Attention is then quantified as:
  (Part 2 Correct Responses + Part 3 Correct Responses + Part 4 Correct Responses) - (Part 2 Incorrect Responses + Part 3 Incorrect Responses + Part 4 Incorrect Responses)
Psychomotor Speed | 60 minutes post-drink consumption
  Measure of how well a subject perceives, attends, responds to visual-perceptual information, and performs motor speed and fine motor coordination. To assess psychomotor speed, participants will complete two tests:
  1. The finger tapping test (FTT), which requires subjects respond by pressing the SPACE BAR with their right index finger as many times as they can in 10 seconds. They do this once for practice, and then there are three test trials. The test is repeated with the left hand; and
  2. The symbol digit coding test (SDC), which consists of serial presentations of screens, each of which contains a bank of eight symbols above eight empty boxes. The participant types in the number on the NUMBER ROW that corresponds to the symbol that is highlighted.
  Psychomotor Speed is then quantified as a singular outcome using data aggregated from these two tests as:
  FTT Right Taps Average + FTT Left Taps Average + SDC Correct Responses
Working Memory | 60 minutes post-drink consumption
  Measure of how well a subject can perceive and attend to symbols using short-term memory processes. Working memory is assessed via completion of the 4-part Continuous Performance Test, which requires the subject to respond to the target stimulus "B" but not to any other letter. Stimuli are presented at random and the subject responds by pressing the SPACE BAR.
  Working memory is assessed as: Part 4 Correct Responses - Part 4 Incorrect Responses
Cognitive Flexibility | 60 minutes post-drink consumption
  Measure of how well subject is able to adapt to rapidly changing and increasingly complex set of directions and/or to manipulate the information. Two tests will be used to assess:
  1. the Shifting Attention Test (SAT), where a square or circle appears at the top of the screen and a square and a circle on the bottom. The figures are either red or blue. The participant is asked to match a bottom figure to the top figure by shape or color with the rules changing at random; and
  2. the Stroop Test, which requires participants to identify the words red, yellow, blue, and green appearing on the screen (part 1), when the color of the word matches what the word says (part 2), or when the color of the word does not match what the word says (part 3).
  Cognitive Flexibility is then quantified as a singular outcome using data aggregated from these two tests as: SAT Correct Responses - SAT Errors - Stroop Commission Errors
Resting Metabolic Rate | 50 minutes post-drink consumption
  Resting metabolic rate (kcal/min) will be quantified from resting, fasted analyses of pulmonary gas exchange.
Resting Respiratory Exchange Ratio | 50 minutes post-drink consumption
  Resting respiratory exchange ratio will be quantified from resting, fasted analyses of pulmonary gas exchange.
Total Mood Disturbance | 105-minutes post-drink consumption
  Total mood disturbance will be quantified using the Profile of Mood State Short Form Questionnaire.
Vigor-Activity | 105-minutes post-drink consumption
  Vigor will be quantified using the Profile of Mood State Short Form
Heart rate | pre-drink consumption, 40-minutes post-drink consumption, 110 minutes post-drink consumption
  Heart rate will be quantified from a standard 3-lead ECG
Blood Pressure | pre-drink consumption, 40 minutes post-drink consumption, 110 minutes post-drink consumption
  Systolic, diastolic, and pulse pressures (mmHg) will be quantified from brachial

OTHER OUTCOMES:
Tension | 105 minutes post-drink consumption
  Tension will be quantified using the Profile of Mood State Short Form Questionnaire.
Fatigue | 105 minutes post-drink consumption
  Fatigue will be quantified using the Profile of Mood State Short Form Questionnaire.
Anger | 105 minutes post-drink consumption
  Anger will be quantified using the Profile of Mood State Short Form Questionnaire.
Confusion | 105 minutes post-drink consumption
  Confusion will be quantified using the Profile of Mood State Short Form Questionnaire.
Friendliness | 105 minutes post-drink consumption
  Friendliness will be quantified using the Profile of Mood State Short Form Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States